CLINICAL TRIAL: NCT01967017
Title: Paracervical Block With Lidocaine as a Modality to Decrease IUD Insertion Related Pain
Brief Title: Study of Local Anesthesia as a Method to Decrease IUD Insertion Related Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding was denied.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00078756
Record Dates: First submitted 2012-12-11; First posted 2013-10-22 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: IUD Insertion Complication; Pain Control
Keywords: Intrauterine device; Paracervical block
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Experimental): Paracervical block using 15 mL of 1 % lidocaine
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): paracervical block using 15 mL of bacteriostatic saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine
  Arms: Lidocaine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Despite the high efficacy of intrauterine devices (IUDs), some women choose not to receive IUDs secondary to the pain associated with insertion. Nulliparous women may be especially susceptible to procedure-related pain from IUD insertion. This study will investigate the difference in perceived pain from IUD insertion, comparing local anesthesia to a placebo, among women who have not had a vaginal delivery before. The investigators anticipate that among women who have not had a previous vaginal delivery, the pain associated with IUD insertion will be significantly decreased after administration of local anesthesia.

DETAILED DESCRIPTION:
The study will investigate the difference in perceived pain from IUD insertion, comparing paracervical block with lidocaine to a placebo (bacteriostatic saline) block, among nulliparous and "functionally nulliparous" women. The investigators plan a double-masked, placebo controlled, randomized clinical trial. The investigators anticipate that among patients who have not had a previous vaginal delivery, the pain associated with IUD insertion will be significantly decreased after administration of a 15 mL 1% lidocaine paracervical block compared to patients who receive 15 mL of bacteriostatic saline (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous and "functionally nulliparous" women receiving their first IUD. "Functionally nulliparous" women include those who have never had a prior vaginal delivery or who have never experienced previous significant cervical dilation (ie. women who have experienced miscarriages or abortions prior to 24 weeks gestation, and women who have had cesarean sections while not in active labor defined as <4 cm dilation).
* English speaking

Exclusion Criteria:

* Presence of a Centers for Disease Control Medical Eligibility Criteria for Contraceptive Use category 3 or 4 precaution to a levonorgestrel IUD
* chronic narcotic use, current or past history of illegal drug use (excluding marijuana)
* allergy to lidocaine

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pain at time of IUD insertion | During IUD insertion (no further follow up after patient leaves ofice)
  Differences in visual analog scale (VAS) measurements of perceived pain at the time of IUD deployment

SECONDARY OUTCOMES:
Pain at other time points of pelvic exam | During other steps of pelvic exam up to 15b minutes after IUD inserted (no further follow up after patient leaves office)
  Intrapersonal and group differences in VAS measurements of expected pain and other time points

OTHER OUTCOMES:
Ease of insertion | Within 15 minutes of IUD insertion
  The degree of difficulty of insertion as rated by the provider will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States